CLINICAL TRIAL: NCT05169567
Title: postMONARCH: A Randomized, Double Blind, Placebo-Controlled, Phase 3 Study to Compare the Efficacy of Abemaciclib Plus Fulvestrant to Placebo Plus Fulvestrant in Participants With HR+, HER2-, Advanced or Metastatic Breast Cancer Following Progression on a CDK4 & 6 Inhibitor and Endocrine Therapy
Brief Title: Abemaciclib (LY2835219) Plus Fulvestrant Compared to Placebo Plus Fulvestrant in Previously Treated Breast Cancer
Acronym: postMONARCH
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18238; I3Y-MC-JPEF (Other: Eli Lilly and Company); 2021-002301-10 (EudraCT Number); 2023-506771-10-00 (Other: EU Trial Number)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2021-12-22; First posted 2021-12-27 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Breast Neoplasm; Neoplasm Metastasis
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — abemaciclib; Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Abemaciclib plus Fulvestrant (Experimental): Abemaciclib 150 milligram (mg) administered orally twice daily (BID) on Days 1 to 28 of a 28-day cycle in combination with fulvestrant 500 mg administered intramuscularly (IM) on Days 1 and 15 of Cycle 1, then on Day 1 of Cycle 2 and beyond. Participants received treatment until discontinuation criteria were met.
  Interventions: Drug: Abemaciclib; Drug: Fulvestrant
- Arm B: Placebo plus Fulvestrant (Active Comparator): Placebo administered orally BID on Days 1 to 28 of a 28-day cycle in combination with fulvestrant 500 mg administered IM on Days 1 and 15 of Cycle 1, then on Day 1 of Cycle 2 and beyond. Participants received treatment until discontinuation criteria were met.
  Interventions: Drug: Fulvestrant; Drug: Placebo

INTERVENTIONS:
Drug: Abemaciclib — Administered orally.
  Arms: Arm A: Abemaciclib plus Fulvestrant
Drug: Fulvestrant — Administered IM.
Drug: Placebo — Administered orally.
  Arms: Arm B: Placebo plus Fulvestrant

SUMMARY:
This study will evaluate the effect of adding abemaciclib to fulvestrant for the treatment of hormone receptor-positive (HR+), human epidermal growth factor receptor 2-negative (HER2-) breast cancer that progressed or recurred after previous treatment with a type of drug known as a CDK4/6 inhibitor and endocrine therapy. Participation could last up to 5 years, depending on how you and your tumor respond.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of HR+, HER2- locally advanced or metastatic breast cancer
* Have radiologic evidence of disease progression or recurrence either

  * On treatment with a CDK4/6 inhibitor with aromatase inhibitor (AI) as initial therapy for advanced disease, or
  * On/after treatment with a CDK4/6 inhibitor plus endocrine therapy (ET) administered as adjuvant therapy for early stage breast cancer
* Must be deemed appropriate for treatment with ET
* If female, have a postmenopausal status by natural or surgical means or by ovarian function suppression
* Have Response Evaluable Criteria in Solid Tumors (RECIST) evaluable disease (measurable disease and/or nonmeasurable disease)
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group scale (Oken et al. 1982)
* Have adequate renal, hematologic, and hepatic organ function
* Must be able to swallow capsules/tablets

Exclusion Criteria:

* Have visceral crisis, lymphangitic spread, or leptomeningeal carcinomatosis
* Have symptomatic or untreated central nervous system metastasis
* Have received any systemic therapy between disease recurrence/progression and study screening
* Have received more than 1 line of therapy for advanced or metastatic disease.
* Have received prior chemotherapy for metastatic breast cancer (MBC)
* Have received prior treatment with fulvestrant, any investigational estrogen receptor (ER)-directed therapy (including selective ER degraders [SERDs] and non-SERDs), any phosphatidylinositol 3-kinase (PI3K)-, mammalian target of rapamycin (mTOR)-, or protein kinase B (AKT)-inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2027-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (138):
- United States (60):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Highlands Oncology Group, Springdale, Arkansas
  - Providence Medical Foundation, Fullerton, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - TRIO-US (Translational Research in Oncology-US), Los Angeles, California
  - Keck School of Medicine of USC, Los Angeles, California
  - UCLA Hematology/Oncology - Parkside, Santa Monica, California
  - Olive View-UCLA Medical Center, Sylmar, California
  - Torrance Memorial Physician Network / Cancer Care, Torrance, California
  - PIH Health Hematology Medical Oncology, Whittier, California
  - Rocky Mountain Cancer Center - Hale Parkway, Denver, Colorado
  - Florida Cancer Specialists SOUTH/Sarah Cannon Research Institute/SCRI, Fort Myers, Florida
  - Millennium Oncology Research Clinic, Hollywood, Florida
  - University of Miami Hospital and Clinics, Sylvester Cancer Center, Miami, Florida
  - Woodlands Medical Specialists, PA, Pensacola, Florida
  - Florida Cancer Specialists SOUTH/Sarah Cannon Research Institute/SCRI, Sarasota, Florida
  - Florida Cancer Specialists EAST/Sarah Cannon Research Institute/SCRI, West Palm Beach, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Central Georgia Cancer Care, Macon, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Hematology Oncology Clinic- Baton Rouge/Sarah Cannon Research Institute/SCRI, Baton Rouge, Louisiana
  - Clinical Trials of SWLA, Lake Charles, Louisiana
  - Central Maine Medical Center, Lewiston, Maine
  - Mfsmc-Hjwci, Baltimore, Maryland
  - Maryland Oncology Hematology, P.A. - Clinton, Clinton, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - MGH Northshore Cancer Center, Danvers, Massachusetts
  - Southcoast Centers for Cancer Care, Fairhaven, Massachusetts
  - Dana-Farber Cancer Institute - Foxborough, Foxborough, Massachusetts
  - Dana Farber Cancer Center Merrimack Valley, Methuen, Massachusetts
  - Dana Farber Cancer Institute, Milford, Massachusetts
  - Mass General Cancer Center, Newton, Massachusetts
  - Dana Farber Cancer Institute, South Weymouth, Massachusetts
  - Reliant Medical Group, Worcester, Massachusetts
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - Dana Farber Cancer Center Londonderry, Londonderry, New Hampshire
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Lifespan Cancer Institute, Providence, Rhode Island
  - Tennessee Oncology-Chattanooga /Sarah Cannon Research Institute/SCRI, Chattanooga, Tennessee
  - Sarah Cannon Research Institute/SCRI, Nashville, Tennessee
  - Tennessee Oncology-Nashville/Sarah Cannon Research Institute/SCRI, Nashville, Tennessee
  - Texas Oncology - Bedford, Bedford, Texas
  - Texas Oncology - Denton, Denton, Texas
  - Texas Oncology, P.A., El Paso, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology - McKinney, McKinney, Texas
  - Woodlands Medical Specialists, PA, McKinney, Texas
  - Woodlands Medical Specialists, PA, Mesquite, Texas
  - Texas Oncology - Plano East, Plano, Texas
  - Texas Oncology-Plano West, Plano, Texas
  - Mays Cancer Center, San Antonio, Texas
  - US Oncology, The Woodlands, Texas
  - Texas Oncology - Tyler Cancer Center, Tyler, Texas
  - Intermountain Medical Center, Murray, Utah
  - Intermountain Healthcare - St. George, St. George, Utah
  - The University of Vermont Medical Center Inc., Burlington, Vermont
  - Shenandoah Oncology, P.C., Winchester, Virginia
- Argentina (6):
  - Fundación Cenit Para La Investigación En Neurociencias, CABA, Buenos Aires F.D.
  - Fundación Respirar, Buenos Aires, Buenos Air
  - Centro de Investigaciones Metabólicas (CINME), Ciudad Autónoma de Buenos Aire, Buenos Air
  - Instituto Médico Río Cuarto, Río Cuarto, Córdoba Province
  - Centro Medico San Roque, San Miguel de Tucumán, Tucumán Province
  - CER San Juan, San Juan
- Belgium (3):
  - Algemeen Ziekenhuis klina, Brasschaat, Antwerpen
  - Jessa Ziekenhuis, Hasselt, Limburg
  - CHU UCL Namur/Site Sainte Elisabeth, Namur
- Czechia (2):
  - Multiscan, Pardubice, Pardubický kraj
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
- Denmark (2):
  - Herlev and Gentofte Hospital, Copenhagen, Capital Region
  - Regionshospitalet Gødstrup, Herning, Central Jutland
- France (4):
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux, Aquitaine
  - CHRU de Brest, Brest, Finistère
  - Hôpital privé du Confluent SAS, Nantes, Loire-Atlantique
  - CHD Vendee, La Roche-sur-Yon, Vendée
- Greece (4):
  - University Hospital of Patras, Pátrai, Achaḯa
  - Alexandra Hospital, Athens, Attikí
  - University General Hospital of Heraklion, Heraklion, Irakleío
  - Euromedica General Clinic of Thessaloniki, Thessaloniki
- Hungary (4):
  - Bacs-Kiskun Megyei Korhaz, Kecskemét, Bács-Kiskun county
  - Petz Aladar Egyetemi Oktato Korhaz, Győr, Győr-Moson-Sopron
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Országos Onkológiai Intézet, Budapest
- Israel (6):
  - Meir Medical Center, Kfar Saba, Central District
  - Rabin Medical Center, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Soroka Medical Center, Beersheba, Southern District
  - Sourasky Medical Center, Tel Aviv, Tell Abīb
- Italy (7):
  - Humanitas Istituto Clinico Catanese, Misterbianco, Catania
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori", Meldola, Emilia-Romagna
  - P.O. "S. Maria della Misericordia" Azienda Sanitaria Universitaria Friuli Centrale, Udine, Friuli Venezia Giulia
  - Instituto Tumori Giovanni Paolo II, Bari
  - Ospedale Misericordia di Grosseto, Grosseto
  - Ospedale San Raffaele, Milan
  - ASL Viterbo Ospedale Belcolle, Viterbo
- Mexico (5):
  - Centro de Investigacion en Artritis y Osteoporosis SC, Mexicali, Estado de Baja California
  - COI Tijuana - Centro Oncológico Internacional, Tijuana, Estado de Baja California
  - Centro Oncológico Internacional (COI), Guadalajara, Jalisco
  - Centro Regiomontano de Investigación, Monterrey, Nuevo León
  - Oncologico Potosino, S.C., San Luis Potosí City, San Luis Potosí
- Poland (2):
  - Europejskie Centrum Zdrowia - Oddzial Onkologii, Otwock, Masovian Voivodeship
  - Opolskie Centrum Onkologii w Opolu im. prof. Tadeusza Koszarowskiego, Opole, Opole Voivodeship
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Korea University Anam Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Korea University Guro Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Kyungpook National University Chilgok Hospital, Daegu, Taegu-Kwangyǒkshi
- Spain (12):
  - CHUAC-Hospital Teresa Herrera, A Coruña, A Coruña [La Coruña]
  - Hospital Universitari Son Espases, Palma, Balears [Baleares]
  - Parc de Salut Mar - Hospital del Mar, Barcelona, Barcelona [Barcelona]
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [Cataluña]
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia, Región de
  - H.R.U Málaga - Hospital Materno-infantil, Málaga, Málaga
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona [Tarragona]
  - Hospital Universitario Doctor Peset, Valencia, Valenciana, Comunitat
  - Hospital Infanta Cristina, Badajoz
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario de Toledo, Toledo
- Sweden (2):
  - Karolinska Universitetssjukhuset Solna, Stockholm, Stockholms
  - Universitetssjukhuset Örebro, Örebro, Örebro Län [se-18]
- Taiwan (6):
  - Chi Mei Medical Center, Tainan, Tainan
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Taipei Tzu Chi General Hospital, New Taipei City
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- Turkey (Türkiye) (9):
  - Izmir Medical Park Hospital, Cordaleo, İzmir
  - Necmettin Erbakan Meram Medical Fac., Meram, Konya
  - Adana City Hospital, Adana
  - Ankara Gülhane Eitim ve Aratrma Hastanesi, Ankara
  - Memorial Ankara Hastanesi, Ankara
  - Dicle Üniversitesi, Diyarbakır
  - Trakya University, Edirne
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul
  - İnönü Üniversitesi Turgut Özal Tıp Merkezi Eğitim ve Araştırma Hastanesi, Malatya

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Zapatero-Solana E, Ding Y, Pulliam N, de Dios A, Ortiz-Ruiz MJ, Lallena MJ. Models of Early Resistance to CDK4/6 Inhibitors Unveil Potential Therapeutic Treatment Sequencing. Int J Mol Sci. 2025 Mar 14;26(6):2643. doi: 10.3390/ijms26062643. PMID 40141282
- [Derived] Kalinsky K, Bianchini G, Hamilton E, Graff SL, Park KH, Jeselsohn R, Demirci U, Martin M, Layman RM, Hurvitz SA, Sammons S, Kaufman PA, Munoz M, Lai JI, Knoderer H, Sandoval C, Chawla AR, Nguyen B, Zhou Y, Ravenberg E, Litchfield LM, Smyth L, Wander SA. Abemaciclib Plus Fulvestrant in Advanced Breast Cancer After Progression on CDK4/6 Inhibition: Results From the Phase III postMONARCH Trial. J Clin Oncol. 2025 Mar 20;43(9):1101-1112. doi: 10.1200/JCO-24-02086. Epub 2024 Dec 18. PMID 39693591
- See also: Abemaciclib (LY2835219) Plus Fulvestrant Compared to Placebo Plus Fulvestrant in Previously Treated Breast Cancer (postMONARCH) — https://trials.lillytrialguide.com/en-US/trial/3dpA0zpCRcFApMyAER3V1o

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers included participants who had an event (progressive disease or death) and participants who were off the treatment and were alive at study conclusion.
Period: Overall Study
Arm/Group | Arm A: Abemaciclib Plus Fulvestrant | Arm B: Placebo Plus Fulvestrant
Started | 182 | 186
Received at Least One Dose of Study Drug | 181 | 185
Completed | 40 | 37
Not Completed | 142 | 149
Not completed — On study treatment | 116 | 128
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 25 | 21

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Arm A: Abemaciclib Plus Fulvestrant: Abemaciclib 150 mg administered orally BID on Days 1 to 28 of a 28-day cycle in combination with fulvestrant 500 mg administered IM on Days 1 and 15 of Cycle 1, then on Day 1 of Cycle 2 and beyond. Participants received treatment until discontinuation criteria were met.
- Total: Total of all reporting groups
Arm/Group | Arm A: Abemaciclib Plus Fulvestrant | Arm B: Placebo Plus Fulvestrant | Total
Number analyzed (Participants) | 182 | 186 | 368
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.00 (12.15) | 59.60 (12.16) | 58.80 (12.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180 | 185 | 365
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 27 | 55
  Not Hispanic or Latino | 135 | 143 | 278
  Unknown or Not Reported | 19 | 16 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 21 | 26 | 47
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 140 | 143 | 283
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 12 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 19 | 20 | 39
  Belgium | 7 | 5 | 12
  Czechia | 1 | 1 | 2
  Denmark | 1 | 2 | 3
  France | 11 | 10 | 21
  Greece | 8 | 4 | 12
  Hungary | 7 | 9 | 16
  Israel | 12 | 11 | 23
  Italy | 16 | 11 | 27
  Mexico | 5 | 4 | 9
  Poland | 2 | 1 | 3
  South Korea | 10 | 10 | 20
  Spain | 27 | 31 | 58
  Taiwan | 11 | 14 | 25
  Turkey | 17 | 25 | 42
  United States | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS defined as the time from the date of randomization to the first evidence of disease progression as defined by response evaluation criteria in solid tumors (RECIST) v1.1 or death from any cause. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. If a participant does not have a complete baseline disease assessment, then the PFS time was censored at the date of randomization, regardless of whether or not objectively determined disease progression or death has been observed for the participant. If a participant was not known to have died or have objective progression as of the data inclusion cutoff date for the analysis, the PFS time was censored at the last adequate tumor assessment date.
Time Frame: Randomization to the date of first documented progression of disease or death from any cause (Up to 21 Months)
Population: All randomized participants (including censored). Censored participants: Abemaciclib plus fulvestrant (n = 65), Placebo plus fulvestrant (n = 45).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Abemaciclib Plus Fulvestrant | Arm B: Placebo Plus Fulvestrant
Number analyzed (Participants) | 182 | 186
Months | 6 [5.6 to 8.1] | 5.3 [3.7 to 5.6]
Statistical Analysis 1: Comparison: Arm A: Abemaciclib Plus Fulvestrant vs Arm B: Placebo Plus Fulvestrant; Test type: Superiority; p = 0.02, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.57 to 0.95]

2. Secondary Outcome: Progression Free Survival (PFS) Determined by Blinded Independent Central Review (BICR)
Description: PFS is defined as the time from the date of randomization to the earliest date of disease progression determined by blinded independent central review (BICR) or death from any cause, whichever occurs first.
Time Frame: Randomization to the date of first documented progression of disease or death from any cause (Up to 22 Months)
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Abemaciclib Plus Fulvestrant | Arm B: Placebo Plus Fulvestrant
Number analyzed (Participants) | 182 | 186
Months | 12.9 [9.5 to NA] — Upper limit of 95% CI was not estimable due to insufficient number of events. | 5.6 [3.9 to 7.7]

3. Secondary Outcome: Objective Response Rate (ORR): Percentage of Participants Who Achieved a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR)
Description: ORR is the best overall tumor response of CR or PR as classified by the investigator according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1). CR is a disappearance of all target and non-target lesions and normalization of tumor marker level. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of non-target lesions or appearance of new lesions.
Time Frame: Randomization until measured progressive disease (Up to 22 Months)
Population: All randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: Abemaciclib Plus Fulvestrant | Arm B: Placebo Plus Fulvestrant
Number analyzed (Participants) | 182 | 186
Percentage of participants | 24 | 10

ADVERSE EVENTS:
Time Frame: Baseline up to 22 months
Description: All participants who received at least one dose of the study drug, regardless of their eligibility for the study.
Arm/Group | Arm A: Abemaciclib Plus Fulvestrant | Arm B: Placebo Plus Fulvestrant
All-Cause Mortality (participants affected / at risk) | 40/181 | 37/185
Serious Adverse Events (participants affected / at risk) | 44/181 | 20/185
Other Adverse Events (participants affected / at risk) | 173/181 | 131/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Abemaciclib Plus Fulvestrant (N=181) | Arm B: Placebo Plus Fulvestrant (N=185)
Anaemia (Blood and lymphatic system disorders) | 2 (4) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 8 (8) | 4 (4)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Abemaciclib Plus Fulvestrant (N=181) | Arm B: Placebo Plus Fulvestrant (N=185)
Anaemia (Blood and lymphatic system disorders) | 63 (87) | 27 (36)
Leukopenia (Blood and lymphatic system disorders) | 32 (48) | 6 (6)
Lymphopenia (Blood and lymphatic system disorders) | 16 (30) | 4 (6)
Neutropenia (Blood and lymphatic system disorders) | 73 (130) | 6 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 33 (47) | 11 (12)
Abdominal pain (Gastrointestinal disorders) | 41 (46) | 30 (40)
Constipation (Gastrointestinal disorders) | 12 (15) | 12 (12)
Diarrhoea (Gastrointestinal disorders) | 135 (307) | 31 (46)
Nausea (Gastrointestinal disorders) | 59 (75) | 34 (43)
Vomiting (Gastrointestinal disorders) | 35 (46) | 11 (13)
Fatigue (General disorders) | 59 (66) | 43 (52)
Oedema peripheral (General disorders) | 10 (10) | 4 (4)
Pyrexia (General disorders) | 12 (13) | 4 (4)
Covid-19 (Infections and infestations) | 14 (15) | 9 (9)
Urinary tract infection (Infections and infestations) | 14 (18) | 4 (4)
Alanine aminotransferase increased (Investigations) | 23 (25) | 19 (25)
Aspartate aminotransferase increased (Investigations) | 27 (34) | 20 (25)
Blood alkaline phosphatase increased (Investigations) | 12 (14) | 12 (14)
Blood creatinine increased (Investigations) | 20 (28) | 4 (4)
Gamma-glutamyltransferase increased (Investigations) | 16 (21) | 12 (13)
Weight decreased (Investigations) | 11 (11) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 33 (40) | 12 (12)
Hypokalaemia (Metabolism and nutrition disorders) | 16 (22) | 4 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (28) | 23 (24)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 17 (19)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 10 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (10) | 13 (15)
Dizziness (Nervous system disorders) | 14 (16) | 13 (14)
Headache (Nervous system disorders) | 16 (17) | 15 (17)
Neuropathy (Nervous system disorders) | 4 (4) | 12 (17)
Insomnia (Psychiatric disorders) | 12 (12) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (25) | 12 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (18) | 6 (7)
Rash (Skin and subcutaneous tissue disorders) | 16 (18) | 7 (7)
Hot flush (Vascular disorders) | 13 (14) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT05169567/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT05169567/SAP_001.pdf